CLINICAL TRIAL: NCT00845390
Title: Patient Expectations After ICD Implantation
Brief Title: Patient Expectations After Implantable-cardioverter Defibrillator (ICD) Implantation
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CHR #08033561
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICD Patients: ICD patients

SUMMARY:
This study will be a qualitative survey to understand the expectations of defibrillator patients with regards to their device. It is unknown what ICD (implantable-cardioverter defibrillator) patients understand about their device and its purpose, thus we will be talking to them about their device. Also, we will be interested in studying their beliefs on how the ICD impacts their life expectancy and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients are eligible for inclusion. We hope to acquire a wide range of ages but are not limited to a specific set.

Exclusion Criteria:

* Non-English speakers will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICD Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Why did you have an ICD implanted? | after ICD implantation

CONTACTS AND LOCATIONS:
Overall Officials: Rita F Redberg, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Arrhythmia and Device Clinic, San Francisco, California, United States